CLINICAL TRIAL: NCT05066568
Title: Effect of Hypnosis Combined With Transcranial Direct Current Stimulation on Pain Perception and Cortical Excitability in Fibromyalgia: A Blinded Randomized Crossover Sham Controlled Clinical Trial
Brief Title: Effect of Hypnosis Combined With Tdcs on Pain Perception and Cortical Excitability in Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 2019-0688
Record Dates: First submitted 2021-08-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Transcranial Direct Current Stimulation; Hypnosis; Fibromyalgia
Keywords: chronic pain; fibromyalgia; hypnotic analgesia; tDCS; DPMS; Cold pressor test
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Hypnosis; RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: Design: Randomized blinded factorial sham controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding: The researcher will receive a device previously programmed by a research assistant. This way the researcher that perform the Transcranial direct current stimulation does not know if it's a active or sham intervention. The subjects will also be blinded to the nature of the stimulation. The subjects will be asked to answer what intervention they think they recieved after each one of the tDCS sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence of interventions starting with tDCS as the first intervention (Other): Week 1 Active tDCS left dorso-lateral prefrontal cortex. F3 anode F4 catode Area of electrodes: 35 cm2 Current intensity: 2mA Stimulation Time: 20min
  Week 2 Rest The subjects will be asked to remain seated and still for 20 minutes.
  Week 3 Hypnotic analgesia suggestion Classic approach. The intervention starts with a induction with suggestions for the subject to focus her attention in a single stimuli, combined with progressive relaxation. After that, direct suggestions are given for comfort and pain reduction.
  Intervention time: 20 minutes
  Week 4 Active tDCS + Hypnotic analgesia suggestion Intervention Time: 20 minutes.
  Week 5 Sham tDCS + Hypnotic analgesia suggestion The sham tDCS will have the same areas of stimulation of the active tDCS, but the device will turn itself out after 30 seconds.
  Intervention time: 20 minutes
  Interventions: Device: Active Tracranial Direct Current Stimulation; Other: Hypnotic analgesia suggestion; Behavioral: Rest; Other: Active tDCS + Hypnotic analgesia suggestion; Other: Sham tDCS + Hypnotic analgesia suggestion
- Sequence of interventions starting with Hypnosis as the first intervention (Other): Week 1 Hypnotic analgesia suggestion Classic approach. The intervention starts with a induction with suggestions for the subject to focus her attention in a single stimuli, combined with progressive relaxation. After that, direct suggestions are given for comfort and pain reduction.
  Intervention time: 20 minutes
  Week 2 Rest The subjects will be asked to remain seated and still for 20 minutes.
  Week 3 Active tDCS left dorso-lateral prefrontal cortex. F3 anode F4 catode Area of electrodes: 35 cm2 Current intensity: 2mA Stimulation Time: 20min
  Week 4 Sham tDCS + Hypnotic analgesia suggestion The sham tDCS will have the same areas of stimulation of the active tDCS, but the device will turn itself out after 30 seconds.
  Intervention time: 20 minutes
  Week 5 Active tDCS + Hypnotic analgesia suggestion Intervention Time: 20 minutes.
  Interventions: Device: Active Tracranial Direct Current Stimulation; Other: Hypnotic analgesia suggestion; Behavioral: Rest; Other: Active tDCS + Hypnotic analgesia suggestion; Other: Sham tDCS + Hypnotic analgesia suggestion

INTERVENTIONS:
Device: Active Tracranial Direct Current Stimulation — Site: dorsolateral prefrontal cortex. F3 anode and F4 catode. Electrode area: 35cm2 Current Intensity: 2mA Stimulation time: 20 min The current ramps up during 30 seconds reaching 2mA, staying this way until the last 30 seconds of stimulation, in wich the current slowly decreases to zero.
  Other Names: a-tDCS
Other: Hypnotic analgesia suggestion — The hypnotic induction protocol was standardized to be applied equally to all subjects. The protocol for hypnotic analgesia begins with an induction with a sequence of suggestions for the subjects to focus their attention on an individual stimulus, associated with progressive relaxation. After that, direct suggestions are given for comfort and pain reduction. The intervention lasts 20 minutes, with 12 minutes of induction and 8 minutes of hypnotic suggestions to reduce pain and leave the trance.
  Other Names: Hypnosis
Behavioral: Rest — The patient is asked to remain seated still for 20 minutes.
Other: Active tDCS + Hypnotic analgesia suggestion — Site: dorsolateral prefrontal cortex. F3 anode and F4 catode. Electrode area: 35cm2 Current Intensity: 2mA Intervention time: 20 min The current ramps up during 30 seconds reaching 2mA, staying this way until the last 30 seconds of stimulation, in wich the current slowly decreases to zero.
  The hypnotic induction protocol was standardized to be applied equally to all subjects. The protocol for hypnotic analgesia begins with an induction with a sequence of suggestions for the subjects to focus their attention on an individual stimulus, associated with progressive relaxation. After that, direct suggestions are given for comfort and pain reduction. The intervention lasts 20 minutes, with 12 minutes of induction and 8 minutes of hypnotic suggestions to reduce pain and leave the trance.
  Other Names: a-tDCS+HS
Other: Sham tDCS + Hypnotic analgesia suggestion — Site: dorsolateral prefrontal cortex. F3 anode and F4 catode. Electrode area: 35cm2 Current Intensity: 0mA Intervention time: 20 min The current is turned off after 30 seconds. The hypnotic induction protocol was standardized to be applied equally to all subjects. The protocol for hypnotic analgesia begins with an induction with a sequence of suggestions for the subjects to focus their attention on an individual stimulus, associated with progressive relaxation. After that, direct suggestions are given for comfort and pain reduction. The intervention lasts 20 minutes, with 12 minutes of induction and 8 minutes of hypnotic suggestions to reduce pain and leave the trance.
  Other Names: s-tDCS+HS

SUMMARY:
Fibromyalgia is a public health condition, which causes great functional disability. Conventional treatment modalities have been shown a very poor therapeutic response, in that most individuals end up becoming poly-medicated and refractory to treatment. Non-pharmacological techniques with promising effects on the syndrome symptoms include both hypnotic analgesia and the transcranial direct-current stimulation (tDCS). Giving the treatment limitations of this syndrome its important to better understand the pain processess in fibromyalgia and treatments effect. This project was developed in order to evaluate the synergistic effect of a hypnotic analgesia suggestion associated with tDCS over pain levels and cortical excitability in individuals with fibromyalgia over a nociceptive stimulation pattern.

DETAILED DESCRIPTION:
Fibromyalgia is a public health condition, which causes great functional disability. Its consequences pervade the personal and social life of the patient, leading to significant impairments in their interpersonal relationships, including work, family and social spheres. The symptoms affect both the physical and emotional abilities. Conventional treatment modalities have been shown a very poor therapeutic response, in that most individuals end up becoming poly-medicated and refractory to treatment. Non-pharmacological techniques with promising effects on the syndrome symptoms include both hypnotic analgesia and the transcranial direct-current stimulation (tDCS). Giving the treatment limitations of this syndrome its important to better understand the pain processess in fibromyalgia and treatments effect. This project was developed in order to evaluate the synergistic effect of a hypnotic analgesia suggestion associated with tDCS over pain levels and cortical excitability in individuals with fibromyalgia over a nociceptive stimulation pattern. It will be performed as a blinded sham controlled cross-over randomized clinical trial. It will be included 20 female subjects diagnosed with fibromyalgia, according to the 2016 revision of the American College of Rheumatologycriteria (2010;2011), ranging in age from 18 to 65 years old, highly susceptible to the hypnosis technique (score ≥ 8) according to the Waterloo-Stanford Scale of Hypnotic Susceptibility (WSGC). They will be allocated in one of two groups, receiving with each cross-over one of the following interventions: A (active-tDCS), B (hypnotic analgesia suggestion), C (Rest), D (active-tDCS + hypnotic analgesia suggestion) and E (sham-tDCS + hypnotic analgesia suggestion). The primary endpoints will be the level of pain, measured by a numerical pain scale (NPS), during nociceptive stimuli induced by the cold pressor test and Short Intracortical Inhibition (SICI). The secondary endpoints will be descent pain modulation system power through the Conditioned Pain Modulation test (CPM - task); and the cortical excitability assessed by Motor Threshold (MT), Motor Evoked Potential (MEP), Cortical Silent Period (CSP) and Short Intracortical Facilitation (SICF) tests during Transcranial Magnetic Stimulation (TMS). The intra and inter-group comparisons will be made by means of two-way ANOVA followed by Bonferroni. A type I error of 5% and type II error of 20%. The present study hypothesizes a synergistic effect of both interventions on pain intensity reported on the Cold Pressor Test, as well as the reduction in the inhibition of cortical excitability level assessed by the TMS, compared to the same measures in an isolated manner.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Literate
* Fibromyalgia diagnosis according to 2016 American College of Rheumatology criteria
* Pain score ≥ 6 in the Numerical Pain Scale during most of the time in the last 3 months.
* Score ≥ 8 /12 in the Waterloo-Stanford Group Hypnotic Susceptibility Scale C

Exclusion Criteria:

* Contraindication to Transcranial Magnetic Stimulation
* Metallic implant in brain
* Medical implants in brain
* Cardiac Pacemaker
* Cochlear implant
* History of drug or alcohol abuse in the last 6 months
* Neurological disorders
* History of head trauma or neurosurgery
* Decompensated systemic diseases
* Chronic inflammatory diseases (lupus, rheumatoid arthritis, Sjogren syndrome, Reiter syndrome)
* Decompensated hypothyroidism
* History of cancer

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain Levels during Cold Pressor Test from Pre to Post Interventions | First assessed 40 minutes Pre interventions and 70 minutes post interventions
  Pain levels measured by a numerical visual analogue scale during Cold Pressor Test. The subject will have her hand submerged in cold water at 0 degrees celcius up to 2 minutes.
Changes in Pain Tolerance during Cold Pressor Test from Pre to Post Interventions | First assessed 40 minutes Pre interventions and again 70 minutes post interventions
  The time in the subject withstands with his hand submerged in cold water at 0 degrees celcius during Cold Pressor Test. With a maximum of 2 minutes.
Changes in Short Cortical Inhibition during Transcranial Magnetic Stimulation from pre to post interventions | First assessed 10 minutes Pre intervention and again 20 minutes post intervention
  Short Cortical Inhibition measured by Transcranial Magnetic Stimulation. Using the MagOption for MagPro R30 and X100 device with electromyography.

SECONDARY OUTCOMES:
Changes in Numerical Pain Scale during Conditioned Pain Modulation-task from Pre to Post Interventions | First assessed 50 minutes pre interventions and again 1 hour post interventions
  Descending pain modulation system assessed by Conditioned Pain Modulation task. The subject will be asked to put her non-dominant hand in a bucket with cold water at 0 degrees celsius. The other forearm will receive a painful heat stimuli using a device. The CPM score is calculated using the difference between the mean pain of both arms during the outcome assessment.
Changes in Motor Threshold from Pre to Post Interventions | First assessed 30 minutes Pre interventions and again immediately post interventions
  Motor Threshold assessed by Transcranial Magnetic Stimulation
Changes in Motor Evoked Potential from Pre to Post Interventions | First assessed 25 minutes Pre interventions and again 5 minutes post interventions
  Motor Evoked Potential assessed by Transcranial Magnetic Stimulation
Changes in Silent Period from Pre to Post Interventions | First assessed 5 minutes Pre Interventions and again 25 minutes post interventions
  Silent Period assessed by Transcranial Magnetic Stimulation
Changes in Intra-cortical Facilitation from Pre to Post Interventions | First assessed 10 minutes Pre intervention and again 20 minutes post intervention
  Intra-cortical Facilitation assessed by Transcranial Magnetic Stimulation

OTHER OUTCOMES:
Pain Catastrophizing Scale | 5 minutes
  Measure of confounding factors
Pittsburgh Sleep Quality Index | 5 minutes
  Measure of confounding factors
Beck Depression Inventory II | 5 minutes
  Measure of confounding factors
State-Trait Anxiety Inventory | 5 minutes
  Measure of confounding factors
Central Sensitization Inventory | 5 minutes
  Measure of confounding factors

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schein B, Beltran G, Franca BR, Sanches PRS, Silva DP Jr, Torres IL, Fegni F, Caumo W. Effects of Hypnotic Analgesia and Transcranial Direct Current Stimulation on Pain Tolerance and Corticospinal Excitability in Individuals with Fibromyalgia: A Cross-Over Randomized Clinical Trial. J Pain Res. 2023 Jan 24;16:187-203. doi: 10.2147/JPR.S384373. eCollection 2023. PMID 36718400